CLINICAL TRIAL: NCT00392691
Title: Ibritumomab Tiuxetan and High-Dose Melphalan as Conditioning Regimen Before Autologous Stem Cell Transplantation for Elderly Patients With Lymphoma in Relapse or Resistant to Chemotherapy. A Multicenter Phase I Trial
Brief Title: Melphalan, Yttrium Y 90 Ibritumomab Tiuxetan, and Rituximab Followed by Autologous Stem Cell Transplant in Treating Older Patients With Non-Hodgkin's Lymphoma That Has Relapsed or Not Responded to Previous Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 37/05; SWS-SAKK-37/05; EU-20648; SPRI-SWS-SAKK-37/05; CDR0000511915
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
Keywords: recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — ibritumomab tiuxetan; Rituximab; Melphalan; Vinorelbine; Granulocyte Colony-Stimulating Factor; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zevalin, Rituximab, Melphalan (Experimental)
  Interventions: Drug: ibritumomab tiuxetan; Drug: rituximab; Drug: melphalan; Drug: vinorelbine tartrate / G-CSF; Procedure: autologous hematopoietic stem cell harvesting and transplantation

INTERVENTIONS:
Drug: ibritumomab tiuxetan — 185 MBq (5mCi) of 111In-Zevalin will be used for radioimaging. and the dose is 14.8 MBq/kg (0.4 mCi/kg) total body weight of 90Y-Zevalin (max. 1184 MBq or 32 mCi at patients > 80kg) for imaging.
  Other Names: ZEVALIN
Drug: rituximab — 250 mg/m2
  Other Names: MabThera
Drug: melphalan — * Dose level 1: 100 mg/m2
  * Dose level 2: 140 mg/m2
  * Dose level 3: 170 mg/m2
  * Dose level 4: 200 mg/m2
  Other Names: Alkeran
Drug: vinorelbine tartrate / G-CSF — on day 1: 35 mg/m2 day 4-8 (longer if required) G-CSF 5 μg/kg s.c. morning and 5 μg/kg s.c. evening for at least 5 days
  Other Names: Navelbine
Procedure: autologous hematopoietic stem cell harvesting and transplantation — Optimal mobilization usually takes place on day 8. A minimum of 2.5x106 CD34+ cells/kg should be collected (optimal 5x106 CD34+ cells/kg). If not enough CD34+ cells can be collected on day 8, it is recommended to continue with G-CSF until a sufficient collection (a minimum of 2.5x106 CD34+ cells/kg) can be obtained.
  Stem cells will be reinfused approximately 24 hours after the melphalan administration. The infusion will be performed with a minimum of 2.5x106 CD34+ cells/kg body weight according to local guidelines. G-CSF (5 μg/kg/d) will be given from day 5 and continued until neutrophils > 0.5x109/l for at least 2 consecutive days.

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as melphalan, before an autologous stem cell transplant helps stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Also, monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan and rituximab, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Chemotherapy and monoclonal antibody therapy also prepares the patient's bone marrow for the stem cell transplant. Giving colony-stimulating factors, such as G-CSF, and vinorelbine helps stem cells move from the bone marrow to the blood so they can be collected and stored. The stem cells are returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and monoclonal antibody therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of melphalan when given together with yttrium Y 90 ibritumomab tiuxetan and rituximab followed by autologous stem cell transplant in treating older patients with non-Hodgkin's lymphoma that has relapsed or not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of high-dose melphalan when given together with yttrium Y 90 ibritumomab tiuxetan and rituximab as a conditioning regimen followed by vinorelbine ditartrate- and filgrastim (G-CSF)-mobilized autologous stem cell transplantation in elderly patients with relapsed or refractory CD20-positive non-Hodgkin's lymphoma.
* Evaluate the feasibility and safety of this regimen in these patients.
* Determine the feasibility of stem cell mobilization with vinorelbine ditartrate in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of high-dose melphalan.

* Stem cell harvest and mobilization: Patients receive vinorelbine ditartrate IV on day -36 and filgrastim (G-CSF) subcutaneously (SC) twice daily on days -33 to -29. Patients undergo peripheral blood stem cell harvest on days -29 to -26.
* Radioimmunotherapy: Patients receive rituximab IV. Within 4 hours after completion of rituximab, patients receive indium In 111 ibritumomab tiuxetan (imaging dose) IV over 10 minutes on day -25. Patients undergo assessment of biodistribution, imaging, and dosimetry on days -25, -22, and optionally on day -20. Patients with acceptable biodistribution of indium In 111 ibritumomab tiuxetan receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan (therapeutic dose) IV over 10 minutes on day -18.
* High-dose chemotherapy: Patients receive high-dose melphalan IV on day -1. Cohorts of 3-6 patients receive escalating doses of high-dose melphalan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
* Autologous stem cell transplantation (ASCT): Patients undergo ASCT on day 0. Patients receive G-CSF SC beginning on day 5 and continuing until blood counts recover.

After completion of study treatment, patients are followed for 100 days.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma of any type
* CD20-positive disease
* Achieved partial or complete response to salvage treatment for relapse or refractory disease within the past 10 weeks
* Must have an indication for autologous stem cell transplantation
* Bone marrow infiltration < 25%
* No evidence of CNS involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* AST ≤ 2 times ULN
* Creatinine clearance > 50 mL/min
* No clinically significant cardiac disease, including any of the following:

  * Unstable angina pectoris
  * Significant arrhythmia
  * Myocardial infarction within the past 3 months
* LVEF > 50%
* No clinically significant urinary tract obstruction
* No clinically significant pulmonary disease
* No serious underlying medical condition that would preclude study participation
* No other malignancy within the past 5 years except nonmelanoma skin cancer or adequately treated in situ cervical cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 30 days since prior participation in another clinical trial
* No prior stem cell transplantation
* No prior radiolabeled antibodies, including for induction of disease remission
* No prior radiotherapy to ≥ 25% of the bone marrow
* No concurrent radiotherapy
* No other concurrent anticancer drugs
* No other concurrent investigational drugs

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of high-dose melphalan in combination with yttrium Y 90 ibritumomab tiuxetan | within 8 weeks after application of melphalan

SECONDARY OUTCOMES:
Toxicity | 100 days (+/- 5 days) after reinfusion of stem cells
Event occurrence up to 100 days after transplantation | up to 100 days after transplantation
Complete remission 100 days after transplantation | 100 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Michele Voegeli, MD, Study Chair — Kantonsspital Liestal; Michele Ghielmini, Prof, Study Chair — IOSI, Ospedale San Giovanni; Angelika Bischof Delaloye, Prof, Study Chair — Faculté de biologie et de médecine de l' Université de Lausanne
Locations (10):
- Switzerland (10):
  - Kantonsspital Aarau, Aarau
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Liestal, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen

REFERENCES:
- [Result] Voegeli M, Rondeau S, Berardi Vilei S, Lerch E, Wannesson L, Pabst T, Rentschler J, Bargetzi M, Jost L, Ketterer N, Bischof Delaloye A, Ghielmini M. Y90 -Ibritumomab tiuxetan (Y90 -IT) and high-dose melphalan as conditioning regimen before autologous stem cell transplantation for elderly patients with lymphoma in relapse or resistant to chemotherapy: a feasibility trial (SAKK 37/05). Hematol Oncol. 2017 Dec;35(4):576-583. doi: 10.1002/hon.2348. Epub 2016 Sep 28. PMID 27677906